CLINICAL TRIAL: NCT05962398
Title: An Extension Study Assessing the Long-term Safety and Efficacy of Etranacogene Dezaparvovec (CSL222) Previously Administered to Adult Male Subjects With Hemophilia B
Brief Title: Long-term Follow-up Study of Male Adults With Hemophilia B Previously Treated With Etranacogene Dezaparvovec (CSL222)
Acronym: IX-TEND 3003
Status: Enrolling by invitation | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: CSL222_3003; EU CT Number (Other: 2023-503765-37-00)
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CSL222: Participants who received CSL222 and completed either the study CSL222_2001 (NCT03489291) or CSL222_3001 (NCT03569891) will be followed up from Year 5 after administration of CSL222 in parent study up to Year 15.
  Interventions: Genetic: AAV5-hFIXco-Padua

INTERVENTIONS:
Genetic: AAV5-hFIXco-Padua — Single intravenous infusion of AAV5-hFIXco-Padua in the study CSL222_2001 (NCT03489291) or CSL222_3001 (NCT03569891).
  Other Names: Etranacogene dezaparvovec

SUMMARY:
The primary purpose of this study is to assess the long-term safety and efficacy in male adults with hemophilia B who were treated with CSL222 (CSL222) in parent studies CSL222_2001 (NCT03489291) or CSL222_3001 (NCT03569891).

ELIGIBILITY:
Inclusion Criteria:

Received treatment with CSL222 in Study CSL222_2001 or Study CSL222_3001, and completed participation in Study CSL222_2001 or Study CSL222_3001 or at least 5 years have passed since receiving CSL222.

Exclusion Criteria:

Not Applicable

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult male participants with hemophilia B who were previously treated with CSL222 in study CSL222_2001 (NCT03489291) or CSL222_3001 (NCT03569891).
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2035-03-23 (Estimated); Study Completion 2035-03-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Serious Adverse Events (SAEs) and AEs of Special Interest (AESIs) | From Year 5 after administration of CSL222 in parent study up to Year 15
Percentage of Participants With SAEs and AESIs | From Year 5 after administration of CSL222 in parent study up to Year 15
Number of SAEs and AESIs | From Year 5 after administration of CSL222 in parent study up to Year 15

SECONDARY OUTCOMES:
Annualized Bleeding Rate (ABR) | From Year 5 after administration of CSL222 in parent study up to Year 15
  The total, spontaneous, joint, and traumatic bleeds will be analyzed.
Number of Participants With Zero Total, Spontaneous, Joint, and Traumatic Bleeding Episodes | From Year 5 after administration of CSL222 in parent study up to Year 15
Endogenous Factor IX (FIX) Activity | From Year 5 after administration of CSL222 in parent study up to Year 15
  Endogenous FIX activity (expressed as percentage [%]) will be assessed using the one-stage activated partial thromboplastin time assay and a chromogenic assay.
Change from Baseline by Visit in Endogenous FIX Activity | At Baseline (in parent study), From Year 5 after administration of CSL222 in parent study up to Year 15
  Endogenous FIX activity (expressed as %) will be assessed using the one-stage activated partial thromboplastin time assay and a chromogenic assay.
Annualized Consumption of FIX Replacement Therapy | From Year 5 after administration of CSL222 in parent study up to Year 15
  The annualized consumption of FIX replacement therapy (excluding FIX replacement for invasive procedures) will be provided.
Annualized Infusion Rate of FIX Replacement Therapy | From Year 5 after administration of CSL222 in parent study up to Year 15
  Annualized infusion rate of FIX replacement therapy (excluding FIX replacement for invasive procedures) will be provided.
Number of Participants Remaining Free of Continuous FIX Prophylaxis | From Year 5 after administration of CSL222 in parent study up to Year 15
Percentage of Participants Remaining Free of Continuous FIX Prophylaxis | From Year 5 after administration of CSL222 in parent study up to Year 15
Number of New Target Joints | From Year 5 after administration of CSL222 in parent study up to Year 15
Percentage Resolution of Pre-existing Target Joints | From Year 5 after administration of CSL222 in parent study up to Year 15
EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Index Value | From Year 5 after administration of CSL222 in parent study up to Year 15
  The EQ-5D-5L questionnaire consists of the EQ-5D-5L descriptive system and the EQ-5D visual analogue scale (VAS). The EQ-5D-5L descriptive system of health-related quality of life (QoL) consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) for which responses will be recorded on 5 levels of severity (no problems, slight problems, moderate problems, severe problems, and extreme problems). The responses will be converted into a single overall health state utility value. This utility value will be derived using the EQ-5D-5L Crosswalk Index Value Calculator v2.xls [Hernández Alava et al, 2023], using the United Kingdom value set.
Change From Baseline in EQ-5D-5L Index Value | Baseline (in parent study), From Year 5 after administration of CSL222 in parent study up to Year 15
  The EQ-5D-5L questionnaire consists of the EQ-5D-5L descriptive system and the EQ-5D VAS. The EQ-5D-5L descriptive system of health-related QoL consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) for which responses will be recorded on 5 levels of severity (no problems, slight problems, moderate problems, severe problems, and extreme problems). The responses will be converted into a single overall health state utility value. This utility value will be derived using the EQ-5D-5L Crosswalk Index Value Calculator v2.xls [Hernández Alava et al, 2023], using the United Kingdom value set.
EQ-5D VAS Score | From Year 5 after administration of CSL222 in parent study up to Year 15
  The EQ-5D VAS, which measures overall health status on a vertical VAS, ranges from 0 to 100. A higher score indicates better QoL.
Change From Baseline in EQ-5D VAS Score | Baseline (in parent study), From Year 5 after administration of CSL222 in parent study up to Year 15
  The EQ-5D VAS, which measures overall health status on a vertical VAS, ranges from 0 to 100. A higher score indicates better QoL.
Hemophilia Quality of Life Questionnaire (Hem-A-QoL) Total Score | From Year 5 after administration of CSL222 in parent study up to Year 15
  The Hem-A-QoL consists of 46 items comprising 10 domains: physical health, feelings, treatment, work and school, dealing with hemophilia, family planning, future, partnerships and sexuality, sports and leisure, and view of yourself for which responses will be recorded from 5 options (never, seldom, sometimes, often, and always; for some items, there is also a "not applicable" option). The total score is based on the scores for each domain and ranges from 0 to 100, with lower scores reflecting a better QoL.
Change From Baseline in Hem-A-QoL Total Score | Baseline (in parent study), From Year 5 after administration of CSL222 in parent study up to Year 15
  The Hem-A-QoL consists of 46 items comprising 10 domains: physical health, feelings, treatment, work and school, dealing with hemophilia, family planning, future, partnerships and sexuality, sports and leisure, and view of yourself for which responses will be recorded from 5 options (never, seldom, sometimes, often, and always; for some items, there is also a "not applicable" option). The total score is based on the scores for each domain and ranges from 0 to 100, with lower scores reflecting a better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (28):
- United States (15):
  - 10-15 Phoenix Childrens Hospital, Phoenix, Arizona
  - 10-14 Arkansas Children's Hospital - Pharmacology, Little Rock, Arkansas
  - 10-22 Orthopaedic Institute for Children, Los Angeles, California
  - 10-21 Children's Hospital of Los Angeles, Los Angeles, California
  - 10-63 UC Davis Medical Center, Sacramento, California
  - 10-12 University of California, San Diego (UCSD), San Diego, California
  - 10-25 University of Colorado Denver, Aurora, Colorado
  - 10-19 University of South Florida, Tampa, Florida
  - 10-10 University of Michigan Medical Center, Ann Arbor, Michigan
  - 10-16 University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - 10-18 Oregon Health & Science University, Portland, Oregon
  - 10-20 Vanderbilt University Medical Center, Nashville, Tennessee
  - 10-28 University of Texas Health Science Center, Houston, Texas
  - 10-26 University of Utah, Salt Lake City, Utah
  - 10-62 Washington Institute for Coagulation, Seattle, Washington
- Belgium (2):
  - 11-31 Cliniques Universitaires Saint-Luc, Brussels
  - 11-30 Universitair Ziekenhuis Leuven, Leuven
- 12-32 Rigshospitalet, Copenhagen, Denmark
- 15-42 Vivantes Klinikum im Friedrichshain - Landsberger Allee, Berlin, Germany
- 19-56 St. James Hospital, Dublin, Ireland
- Netherlands (4):
  - 13-33 Amsterdam Universitair Medische Centra (UMC), Amsterdam-Zuidoost
  - 13-35 University Medical Center Groningen, Groningen
  - 13-34 Erasmus University Medical Center, Rotterdam
  - 13-36 Universitair Medisch Centrum Utrecht, Utrecht
- 16-43 Skane University Hospital, Malmo, Sweden
- United Kingdom (3):
  - 18-52 Barts Health NHS Trust, London, England
  - 18-54 Addenbrooke's Hospital, Cambridge
  - 18-53 University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.

REFERENCES:
- [Derived] von Drygalski A, Gomez E, Giermasz A, Castaman G, Key NS, Lattimore SU, Leebeek FWG, Miesbach WA, Recht M, Monahan PE, Le Quellec S, Pipe SW. Completion of phase 2b trial of etranacogene dezaparvovec gene therapy in patients with hemophilia B over 5 years. Blood Adv. 2025 Jul 22;9(14):3543-3552. doi: 10.1182/bloodadvances.2024015291. PMID 40188458